CLINICAL TRIAL: NCT06674330
Title: National Taiwan University Hospital Yun_Lin Branch
Brief Title: Using a Population Pharmacokinetic Model to Estimate the Dosage of Teicoplanin in Patients With Hematologic Malignancy or Critical Illness
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202406020RIND
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Hematological Malignancies; Critical Illness
Keywords: Model-Informed Precision Dosing; teicoplanin; population pharmacokinetic model
MeSH Terms: conditions — Hematologic Neoplasms; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Months
Biospecimen Retention: Samples Without DNA — Blood sample of patients prescribed with teicoplanin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: concentration of teicoplanin — post analysis of concentration of teicoplanin

SUMMARY:
Model Informed Precision Dosing (MIPD) integrates clinical data to optimize dosing for patients with unstable pharmacokinetics, like those with hematologic malignancies or critical illnesses. This study aims to create a pharmacokinetic model for teicoplanin, addressing complex dosing challenges and improving therapeutic outcomes through MIPD-driven recommendations.

DETAILED DESCRIPTION:
In recent years, there has been a trend towards not only monitoring drug concentrations but also incorporating clinically significant data into mathematical models to provide recommended dosages with improvement of clinical treatment outcomes, known as Model Informed Precision Dosing (MIPD). The purpose of MIPD is to address the challenges faced by patients with unstable pharmacokinetics, such as those with hematologic malignancies or critical illnesses. These patients often struggle to achieve stable drug concentrations due to various factors, leading to suboptimal therapeutic effects. Both hematologic malignancy and critically ill patients are prone to infections. Since pathogens are difficult to diagnose early, the primary strategy is to administer broad-spectrum antibiotics that cover Gram-positive bacterial infections. Teicoplanin, a glycopeptide antibiotic, is used to treat infections caused by Gram-positive bacteria, including Staphylococcus aureus. However, due to its long elimination half-life (83~182 hours), It has been a clinical challenge to determine the appropriate dosage. Additionally, these two patient groups often exhibit hypoalbuminemia and unstable renal function. Since teicoplanin is highly protein-bound (90-95% bound) and primarily excreted by the kidneys (97% excretion), optimal dosing recommendations require therapeutic monitoring to achieve better treatment outcomes.

Recommended target of therapeutic drug monitoring was established by the Japanese Society of Infectious Diseases in 2022. The targeted pharmacokinetic pharmacodynamic parameter is the 24 hours area under the curve to minimum inhibitory concentration (AUC24/MIC). Since MIPD software to estimate AUC of teicoplanin is not available in many institutions, achieving the trough level target is recommended. Our previous study found that, following a loading dose regimen of 12 mg/kg/dose every 12 hours for three doses, followed by a fourth dose at the 24th hour, hematologic malignancy patients achieved the best therapeutic effect if the trough level reached ≥18.85 mcg/ml at 48 hours.

This research aims to retrospectively construct a population pharmacokinetic model by using data from hematologic malignancy patients. Moreover, it will prospectively apply MIPD concept to provide optimal clinical dosage recommendations for hematologic malignancy or critically ill patients and subsequently analyzing the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged over 20 diagnosed with hematologic malignancy or critical illness.
* Clinically require teicoplanin for treating fever with suspected Gram-positive bacterial infection for more than 48 hours.

Exclusion Criteria:

* Adult patients without hematologic malignancy or critical illness.
* Patients not using teicoplanin for fever with suspected Gram-positive bacterial infection.
* patients receiving renal dialysis within 48 hours of starting teicoplanin.
* Patients treated with teicoplanin for less than 48 hours.
* Pregnant women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Hematologic Malignancy Group: Patients with cancers affecting blood, bone marrow, or lymph nodes, such as leukemia or lymphoma.
  * Critical Illness Group: Patients with life-threatening conditions requiring intensive care, often with unstable vital signs or organ dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
use population pharmacokinetics model to find out the risk factors | From enrollment to the end of treatment at last 2 weeks

IPD SHARING:
Plan to Share IPD: No